CLINICAL TRIAL: NCT05965297
Title: Comparison of Two Conventional Glass Ionomer Cements in the Restoration of Posterior Class II Lesion in the Primary Dentition: a Randomized Controlled Non Inferiority Trial
Brief Title: Comparison of Two GIC's in the Restoration of Posterior Class II Lesions in the Primary Dentition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Collaborators: University of Coimbra (Other); University Arthur Sá Earp Neto (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DeltaFill
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Dental Caries
Keywords: Primary Dentition; Glass ionomer cements; Posterior Class II restorations; DeltaFil; Riva Self Cure HV
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Noninferiority trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DeltaFil (Experimental): Class II restorations are placed in primary molars after conventional cavity preparation.
  Interventions: Device: DeltaFil
- Riva Self Cure HV (Active Comparator): Class II restorations are placed in primary molars after conventional cavity preparation.
  Interventions: Device: Riva Self Cure HV

INTERVENTIONS:
Device: DeltaFil — Cavities are prepared using rotary instruments/diamond burs. Afterwards, the cavity is conditioned (using DeltaFil conditioner) and cleaned, with subsequent insertion of a conventional restorative glass-ionomer (DeltaFil). During the curing phase and after finishing Riva Coat will be applied to all restoration surfaces for moisture protection.
  Arms: DeltaFil
Device: Riva Self Cure HV — Cavities are prepared using rotary instruments/diamond burs. Afterwards, the cavity is conditioned (using Riva conditioner) and cleaned, with subsequent insertion of a conventional restorative glass-ionomer (Riva Self Cure HV). During the curing phase and after finishing Riva Coat will be applied to all restoration surfaces for moisture protection.
  Arms: Riva Self Cure HV

SUMMARY:
This study will investigate the clinical performance of a novel restorative glass ionomer (DeltaFil, DMG) in comparison to an established restorative glass ionomer (Riva Self Cure HV, SDI) in the restoration of Class II cavities in primary molars.

DETAILED DESCRIPTION:
Dental caries (tooth decay) remains one of the most prevalent diseases worldwide. It is a dynamic and continuous process that, if uncontrolled, eventually leads to cavitation and the need for restorative treatment to maintain the form and function of the tooth.Today there are many possibilities for direct restorations, e.g. resin composites, compomers, resin-modified glass ionomer cements (RMGICs) and glass ionomer cements (GICs), which all offer their own advantages and disadvantages.

GIC are particularly suitable for treatments in young patients due to their high biocompatibility, fluoride release, less moisture and technique sensitivity as well as compatibility with Atraumatic restorative treatment (ART) treatment. However, these materials have lower mechanical properties compared to other restorative materials, which negatively affects the survival rate when placed in load bearing areas. Fracture, loss and wear being the most common causes for failure.

This randomized, controlled non-inferiority trial aims to evaluate the performance of the new restorative glass ionomer DeltaFil, that offers an increased fracture toughness, in comparison to an established restorative glass-ionomer (Riva Self Cure HV).

ELIGIBILITY:
Inclusion Criteria:

* At least 1 and up to 3 primary molars with either International Caries Detection and Assessment System (ICDAS) lesions stage 2-5 or preexisting restorations requiring placement/replacement of Class II restorations
* Defects limited to occlusal-proximal surface, with cavity sizes smaller than 3 mm mesio-distally and 3 mm in the occluso-cervical and bucco-lingual directions measured with a World Health Organization (WHO)-graded periodontal probe
* Teeth should have both adjoining and their antagonist teeth present. After restoration the restored tooth should enable appropriate proximal contacts on both mesial and distal surfaces after setting of the class II restoration and be in occlusion with the antagonist tooth
* Good access
* Good general health (ASA I, II)
* Good oral hygiene (OHI-S < 1.9)
* Guardians have given informed consent
* Child is cooperative and assented

Exclusion Criteria:

* Known allergy/ sensitivity to GIC or other materials used in this study
* Space maintainers or orthodontic appliances
* Tooth has a caries lesion or restoration other than those included in the study
* Tooth has pathological mobility
* Tooth has preexisting developmental defects
* Tooth with pulp exposure or indication for endodontic treatment
* Pain, fistula or abscess related to the selected tooth
* Obvious signs of parafunctional habits (e.g. bruxism)
* Participation in another study
* Incapable to participate in the recall visits at the university hospital

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Survival rate of Class II restorations | 24 months
  Restorations are clinically assessed using the Fédération Dentaire Internationale (FDI) criteria. A "surviving" restoration is defined as a restoration that is still present at the time of evaluation and has no individual FDI criteria with a score of 5 (clinically poor).

SECONDARY OUTCOMES:
Survival rate of Class II restorations | 6, 12, 36, 48 and 60 months
  Restorations are clinically assessed using the FDI criteria. A "surviving" restoration is defined as a restoration that is still present at the time of evaluation and has no individual FDI criteria with a score of 5 (clinically poor).
Individual FDI parameter assessment | Baseline, 6, 12, 24, 36, 48 and 60 months
  Restorations are clinically assessed using the FDI criteria. Specifically, the following criteria are assessed individually on a scale from 1 "very good" to 5 "clinicially poor":
  Esthetic properties (Surface Luster; Surface Staining; Color Match; Anatomical Form); Functional properties (Fractures and Retention; Wear; Approximal Contact Point and Contour; Patient view); Biological properties (Postoperative Hypersensitivity & Tooth Vitality; Recurrence of Caries, Erosion, Abfraction; Periodontal Response; Tooth Integrity;Adjacent mucosa)

OTHER OUTCOMES:
Caries Experience | Baseline, 6, 12, 24, 36, 48 and 60 months
  To assess caries experience the dmft score will be recorded. dmft refers to the number of primary teeth (t) with either decay (d), missing due to caries (m) or a filling (f).
Oral Hygiene | Baseline, 6, 12, 24, 36, 48 and 60 months
  Oral hygiene will be assessed using the Oral Hygiene Index-Simplified (OHI-S).

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Effenberger, Dr., Study Chair — DMG Dental Material Gesellschaft mbH
Locations (2):
- University Arthur Sá Earp Neto, Dental School - Pediatric Dentistry Clinic, Petrópolis, Brazil
- University of Coimbra, Faculty of Medicine, Paediatric and Preventive Dentistry Institute, Coimbra, Portugal

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774